CLINICAL TRIAL: NCT04797429
Title: Improving Glycaemic Control in Patients With Type 2 Diabetes Mellitus Through Peer Support Instant Messaging: a Randomized Controlled Trial
Brief Title: Improving Glycaemic Control in Patients With Type 2 Diabetes Mellitus Through Peer Support Instant Messaging
Acronym: DiabPeerS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Pölten University of Applied Sciences (Other)
Collaborators: Karl Landsteiner University of Health Sciences (Other); Austrian Health Insurance Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LS18-021
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Peer Support; Instant Messaging Service
Keywords: Diabetes Mellitus Type 2; Online Intervention; Peer Support; Instant Messaging Service; Glycaemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: blinding is not possible because of obvious differences between the interventions: the intervention group participates in the IMS-intervention and the control group does not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will receive antidiabetic therapy according to the current guidelines but with the additional opportunity to use the peer support IMS tool. Peer support and moderation of the intervention group will be provided by moderators. Moderators will be supervised by a dietitian.
  Interventions: Other: Peer Support Intervention via Instant Messaging Service Tool (IMS-Tool)
- control group (Active Comparator): The control group receives the antidiabetic therapy according to the current guidelines, but without having access to the IMS tool. This means that participants receive medical treatment by their practitioner according to the Austrian recommendations.
  Interventions: Other: antidiabetic therapy according to the current guidelines

INTERVENTIONS:
Other: Peer Support Intervention via Instant Messaging Service Tool (IMS-Tool) — Peer Support via the IMS-tool increases diabetes self-management, improves self-efficiacy, adherence and glycaemic control
  Arms: intervention group
Other: antidiabetic therapy according to the current guidelines — In contrast, the control group has to manage their diabetes mellitus type 2 with standard support and without online exchange.
  Arms: control group

SUMMARY:
Diabetes mellitus is one of the four priority non-communicable diseases worldwide. Globally, 425 million adults suffered from diabetes mellitus (7.2-11.3%) in 2017 and the International Diabetes Federation estimates an increase of 48% of the prevalence until 2045. Type 2 diabetes, which is the most common type of diabetes, is mainly seen in adults older than 40 years. Diabetes can lead to serious long-term complications as well as a lower quality of life, worse mental health, and a reduced life expectancy. Due to the chronical character of diabetes, the disease requires continuous therapy, regular medical appointments, and good adherence of those suffering. Therefore, diabetes self-management education (DSME) plays a significant role to increase patient's self-management capacity and improve diabetes therapy. Research indicates that these outcomes might be difficult to maintain and seem to decline soon after DSME ends. Consequently, effective strategies to preserve the positive effects of DSME are needed. Preliminary results show that peer support, which means support from a person who has experiential knowledge of a specific behaviour or stressor and similar characteristics as the target population, is associated with better outcomes in terms of HbA1c, cardiovascular disease risk factors or self-efficacy at lower cost compared to standard therapy. Although those results are promising, research on peer support in diabetes care is still in its infancy and the influence of various factors is unclear. Peer support instant messaging services (IMS) approaches have significant potential for diabetes management because support can be provided easily and prompt, is inexpensive, and needs less effort to attend compared to standard therapy. Furthermore, almost half of the 40-69-year-old age group, which is mostly affected by the onset of type 2 diabetes, use IMS. The major objective of the project is to analyse the impact of a peer supported IMS intervention in addition to a standard diabetes therapy on the glycaemic control of type 2 diabetic patients. A total of 205 participants (196 participants and 9 moderators) with type 2 diabetes mellitus, older than 40 years will be included and randomly assigned to the intervention or control group. Both groups will receive standard therapy, but the intervention group will use the peer support IMS tool, additionally. The duration of the intervention will last for seven months, followed by a follow-up of seven months. Biochemical, behavioural, and psychosocial parameters will be measured before, in the middle, and after the intervention as well as after the follow-up.

ELIGIBILITY:
Inclusion criteria participants exclusive moderators:

* diagnosed type 2 diabetes mellitus according to the Austrian definition
* HbA1c of ≥ 6.5% (48 mmol/mol) at the last measurement
* receive the antidiabetic therapy according to the current guidelines
* older than 40 years
* living in Lower Austria
* get oral hyperglycaemic agents for maximum three years
* understand the individual commitments during trial
* must be able to visit training and measurements

Inclusion criteria moderators:

* diagnosed type 2 diabetes mellitus according to the Austrian definition
* HbA1c of ≥ 6.5% (48 mmol/mol) at the last measurement
* receive the antidiabetic therapy according to the current guidelines
* get oral hyperglycaemic agents for three years minimum
* older than 60 years
* living in the vicinity of the training location in St. Pölten, which means residing in St. Pölten, St. Pölten Land, Melk, Krems, or Lilienfeld
* engaged participating (= regular participation) in the Austrian disease management program 'Therapie aktiv - Diabetes im Griff'
* understand the individual commitments during trial
* must be able to visit training and measurements
* commitment to undergo the moderator training

Exclusion Criteria for all participants:

* hospitalization of more than 3 weeks during the intervention
* eye disorders that severely limit vision and, hence, inability to read the display (e.g., proliferative retinopathy or macular edema)
* severe illnesses such as kidney, liver, heart disease, or malignant cancer, neurological of mental illness which make a longer hospitalization likely
* substance abuse
* pregnancy
* limitation in the German language
* unable to visit training and measurements

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
HbA1c [%] (change over a period of 7 months intervention and 7 months follow-up with 4 measurement dates) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  HbA1c = glycated haemoglobin reflects average plasma glucose over the previous 8-12 weeks. It can be tested at any time of the day and does not require special preparation like fasting

SECONDARY OUTCOMES:
Quality of life measured by Short-Form-Health Survey (SF-12) (change over a period of 7 months intervention and 7 months follow-up with 4 measurement dates) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  Quality of life will be measured using the 'Short-Form-Health Survey' (SF-12): the SF-12 includes eight dimensions ('physical functioning', 'role limitations due to physical problems', 'bodily pain', 'vitality', 'general health perceptions' , 'social functioning', 'role limitations due to emotional problems', 'mental health'). The summary scores 'physical component summary' and 'mental component summary' (0-100 scales) can be calculated from the specified scales.
Medication adherence measured by A-14 (change over a period of 7 months intervention and 7 months follow-up with 4 measurement dates) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  Medication adherence will be measured using the 'A14-scale': the A14 consists of 14 items of non-adherent behaviors phrased in a non-threatening and non-judgemental way using a five-item Likert scale with the endpoints '4' (never) to '0' (very often).
Diabetes self-management behaviors measured by 'Summary of Diabetes Self-Care Activities German' (SDSCA-G) (change over a period of 7 months intervention and 7 months follow-up with 4 measurement dates) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  Diabetes self-management behaviors will be measured using the 'Summary of Diabetes Self-Care Activities German' (SDSCA-G): the SDSCA-G focuses on the past seven days related to the diabetes self-care activities 'nutrition', 'physical activities', 'blood glucose testing', 'foot care', and 'smoking'.
Diabetes knowledge will be measured using the 'Diabetes Knowledge Test' (DKT) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  DKT consists of 20 statements about diabetes which have to be rated as 'true', 'false' or 'don't know'. Based on the answers, a difficulty index (percent of patients who scored correctly) is calculated.
Diabetes distress will be measure using the 'Diabetes Distress Scale' (DDS) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  the DDS includes for dimensions of distress ('emotional burden', 'regimen distress', 'interpersonal distress', 'physician distress'). The DDS consists of 17 items using a six-point Likert scale with the endpoints '1' (not a problem) and '5' (a very serious problem).
Depression will be measured using the 'Patient Health Questionnaire-9' (PHQ-9) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  PHQ-9 asks for all nine criteria of depression as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) using a four-point Likert scale with the endpoints '0' (not at all) and '3' (nearly every day).
Social support will be measured using the 'Fragebogen zur Sozialen Unterstützung' (F-SozU) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  F-SozU operationalizes social support as perceived or anticipated support from the social environment. The short form consists of the following subscales: 'emotional support', 'practical support', 'social integration', 'stress from the social network'. The F-SozU involves of 14 items using a five-point Likert scale with the endpoints '1' (does not apply) and '5' (accurate).
Dietary behaviour will be measured using a Food Frequency Questionnaire | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  Asses the dietary behaviour during the last month
Physical activity will be measured using the 'International Physical Activity Questionnaire Short Form' (IPAQ-SF) | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  IPAQ-SF asks seven questions to assess 'vigorous-intensity' and 'moderate-intensity' physical activity as well as 'walking' and 'sitting'. Participants indicate the time in minutes or hours for each activity level. Based on this information, three levels of physical activity (low, moderate, high) are calculated and expressed in metabolic equivalent of task (MET) minutes per week.
Biochemical parameters | at baseline, three months after the start of the intervention, at the end of the intervention = seven months after the start of the intervention, follow-up = 14 months after the start of the intervention
  fasting blood glucose [mg/dl], total cholesterol [mg/dl], high-density lipoprotein [mg/dl], low-density lipoprotein [mg/dl], blood pressurge [mmHg], body height [cm], body weight [cm], body fat [%]

CONTACTS AND LOCATIONS:
Locations (1):
- Sankt Pölten University of Applied Sciences, Sankt Pölten, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hold E, Grublbauer J, Wiesholzer M, Wewerka-Kreimel D, Stieger S, Kuschei W, Kisser P, Gutzer E, Hemetek U, Ebner-Zarl A, Pripfl J. Improving glycemic control in patients with type 2 diabetes mellitus through a peer support instant messaging service intervention (DiabPeerS): study protocol for a randomized controlled trial. Trials. 2022 Apr 14;23(1):308. doi: 10.1186/s13063-022-06202-2. PMID 35422003